CLINICAL TRIAL: NCT06201962
Title: Effect of Massage and Foot Reflexology on Newborns' Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ayşe Belpınar, Lecturer, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ABozokU
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Preterm Infants; Sleep
Keywords: Preterm Infants; Sleep Wake Cycle; Massage; Foot Reflexology
MeSH Terms: interventions — Massage

STUDY DESIGN:
Intervention Model Description: This study used a randomized controlled trial. A parallel trial design was used describing two different experimental groups (Massage and Foot Reflexology) and a control group
Who Masked: Participant
Masking Description: Because of the nature of the intervention, double-blinding was not possible in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Massage (Experimental): Before the procedure, written and verbal consent will be obtained from the newborn's guardian and brief information will be given about the massage to be performed on the newborn. Before applying massage to premature babies, their 24-hour sleep duration will be evaluated with an actigraphy device. Starting from the face with gentle touches, massage will be applied to the baby's forehead, around the eyes and cheeks with 2 fingers, without pressing too much. Then, the chest area will be massaged with circular movements from right to left, and then the upper and lower extremities will be massaged. Finally, the massage will be completed by turning the baby face down and applying gentle pressure to the back area. Massage applications will be performed for 15 minutes every morning and evening for two days. On the morning of the second day, an actigraphy device will be attached to the premature babies' ankles and their 24-hour sleep will be re-evaluated.
  Interventions: Other: Massage
- Foot Reflexology (Experimental): Before the procedure, written and verbal consent will be obtained from the newborn's guardian and brief information will be given about the foot reflexology to be performed on the newborn. In addition to daily routine nursing care and monitoring for premature babies, before applying foot reflexology, the actigraphy device will be attached to the babies' ankles and their 24-hour sleep duration will be evaluated. In the reflexology group, the researcher will hold the baby's foot with his left hand and gently massage each foot with the thumb of his right hand for 15 minutes. Foot reflexology will be performed for 15 minutes every morning and evening for two days. On the morning of the second day, an actigraphy device will be attached to the premature babies' ankles and their 24-hour sleep will be re-evaluated.
  Interventions: Other: Foot Reflexology
- Control (Experimental): Newborns will receive routine medical treatment and nursing care and will not undergo any procedures. Before the procedure, written and verbal consent will be obtained from the newborn's guardian and brief information about the study will be given. Premature babies will have their 24-hour sleep recorded with actigraphy 1 day in advance. Then, the nursing care that premature babies receive in their daily routine will be given for two days. On the morning of the second day, an actigraphy device will be attached to the left foot of the premature babies and their 24-hour sleep on the second day will be recorded.
  Interventions: Other: Control

INTERVENTIONS:
Other: Massage — Massage applications will be performed for 15 minutes every morning and evening for two days.
  Arms: Massage
Other: Foot Reflexology — In the reflexology group, the researcher will hold the baby's foot with his left hand and gently massage each foot with the thumb of his right hand for 15 minutes.
  Arms: Foot Reflexology
Other: Control — Newborns will receive routine medical treatment and nursing care and will not undergo any procedures.
  Arms: Control

SUMMARY:
Purpose: Newborns undergo biochemical and physiological changes involving all their systems in the first days of their lives and may experience difficulties in adapting to extrauterine life for various reasons. Leaving the warm, dark, quiet, calm, fluid-filled mother's womb of newborns whose systems are not yet mature and placing them in the intensive care unit with many stimuli creates intense stress and negatively affects the sleep-wake pattern required for growth-development and neurodevelopment. It is intensive for the development of newborns' neurosensory systems. They have sleep requirements. It is known that the brain activity of newborns during the intrauterine period is similar to REM (Rapid Eye Movement) sleep activity, they sleep more than adults, and they spend most of their sleep in the REM sleep period. For this reason, our research will be conducted to examine the effects of massage and foot reflexology applied to preterm newborns on sleep.

Design and Methods: This randomized experimental study was carried out on 108 preterm newborns with gestational weeks between 30-37, hospitalized in the neonatal intensive care unit of a city hospital. The researcher was applied massage (n:36) and foot reflexology (n:36) to the newborns for 15 minutes, twice a day for 2 days. No intervention other than routine clinical practices was applied to the control group (n:36). The 24-hour sleep of the newborns included in the study was monitored with a sleep-wakefulness measuring device before the application and on the day the naps end, and was recorded in the newborn follow-up form. Statistical analysis was performed using percentages, means, median, variance and Kruskal Wallis, Wilcoxon tests test.

DETAILED DESCRIPTION:
Sleep is very important for human life and developmentally involves both physiological and mental processes. Sleep is considered not only as a state of rest, but also as a state of intense brain development in which neurotransmitters specific to each sleep stage affect brain maturation . Newborns sleep an average of 16-20 hours a day, spending most of their sleep in the REM (Rapid Eye Movement Phase) sleep period. For this reason, sleep quality in the neonatal period directly affects healthy growth and development. Newborns, who leave the warm, dark, quiet, calm, amniotic fluid-filled mother's womb at birth, undergo biochemical and physiological changes involving all their systems in the first days of their lives and may experience difficulties in adapting to extrauterine life due to various reasons .

Babies who leave the intrauterine period early are admitted to technologically equipped neonatal intensive care units. In the neonatal intensive care unit, they are exposed to many stressful stimuli and environmental factors. Premature babies are exposed to painful invasive procedures in the neonatal intensive care unit, negative environmental conditions such as frequent feeding, exposure to high-frequency sounds and constant light negatively affect their sleep-wake cycles.

There are studies in the literature to determine the sleep and wakefulness status of premature babies and the factors affecting them. There are studies examining massage, position and music practices applied to preterm babies. It was observed that the number of babies sleeping was higher in the measurements made after massage therapy in premature babies who received massage and premature babies who did not. Additionally, in his systematic review of massage practice; It has been revealed that it increases mother-baby interaction and positively affects sleep conditions by reducing stress levels and crying .

Today, the use of complementary and alternative medicine treatments is increasing in healthcare systems all over the world. Nurses can use these ways, along with regular treatments, to improve health. In this context, foot reflexology, one of the six most commonly used treatments in complementary medicine, is effective not only in the treatment of diseases but also in protecting health. Reflexology is defined as the science that stimulates the ends of sensory nerves connected to receptors and points related to the internal organs of the body using different degrees of pressure, such as massage and touch. By applying the compression technique to the reflection point of each organ using reflexology, the blockage in the energy flow path is removed and as a result, the energy flows in the movement channels. It has been stated that foot reflexology can improve the physiological index and reduce O2 saturation, heart rate, and inspire relaxation in newborns . There are studies examining the effects of invasive procedures on pain, comfort and physiological parameters .

Developing individualized supportive interventions that ensure deep sleep and wakefulness is important for the quality of care provided to preterm infants. For this reason, it is important to reduce the negativities caused by neonatal intensive care units, improve care, reduce pain caused by invasive procedures and the environment, and ensure the sleep quality and order of premature babies.

There are studies in the literature about the effects of massage and foot reflexology on pain, comfort and vital signs in preterm babies, but no study has been found comparing these methods and examining their effects on sleep. In the literature review, while there are studies in which parents subjectively evaluate children's sleep, no other studies were found in which premature babies' sleep is measured objectively. Therefore, it will be carried out to examine the effects of massage and foot reflexology applied to premature babies on sleep.

ELIGIBILITY:
Inclusion Criteria:

* Those born between 30-37 weeks of gestation and hospitalized in the Neonatal Intensive Care Unit

  * Those who have a healthy skin structure (no acne, urticaria, eczema or any allergic problems)
  * Birth weight of 1500 g and above,
  * Do not have a medical condition (surgical intervention, mass, umbilical catheter, etc.) that contraindicates area massage.
  * Those whose vital signs are stable

Exclusion Criteria:

* Those whose vital signs are stable
* Those with foot anomalies or those who underwent outpatient surgery
* Those dependent on high-frequency mechanical ventilation
* Those receiving sedative treatment
* Those with hyperbilirubinemia
* Babies with hypoglycemia or hyperglycemia
* Those with genetic and congenital anomalies

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Preterm babies will be included in each group in equal numbers as boys and girls.
Enrollment: 108 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Changes in sleep | 24 hours
  The researcher will monitor the newborn babies' sleep times with a sleep-wake measurement device for 24 hours and record them in the Newborn Follow-up Form.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Belpınar, Phd, Principal Investigator — Bozok University
Locations (1):
- Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Groot ER, Knoop MS, van den Hoogen A, Wang X, Long X, Pillen S, Benders M, Dudink J. The value of cardiorespiratory parameters for sleep state classification in preterm infants: A systematic review. Sleep Med Rev. 2021 Aug;58:101462. doi: 10.1016/j.smrv.2021.101462. Epub 2021 Mar 14. PMID 33826975
- [Background] Sentner T, Wang X, de Groot ER, van Schaijk L, Tataranno ML, Vijlbrief DC, Benders MJNL, Bartels R, Dudink J. The Sleep Well Baby project: an automated real-time sleep-wake state prediction algorithm in preterm infants. Sleep. 2022 Oct 10;45(10):zsac143. doi: 10.1093/sleep/zsac143. PMID 35749799
- [Background] Firmino C, Rodrigues M, Franco S, Ferreira J, Simoes AR, Castro C, Fernandes JB. Nursing Interventions That Promote Sleep in Preterm Newborns in the Neonatal Intensive Care Units: An Integrative Review. Int J Environ Res Public Health. 2022 Sep 2;19(17):10953. doi: 10.3390/ijerph191710953. PMID 36078666
- [Background] Park J. Sleep Promotion for Preterm Infants in the NICU. Nurs Womens Health. 2020 Feb;24(1):24-35. doi: 10.1016/j.nwh.2019.11.004. Epub 2020 Feb 19. PMID 32083554
- [Background] Uchitel J, Vanhatalo S, Austin T. Early development of sleep and brain functional connectivity in term-born and preterm infants. Pediatr Res. 2022 Mar;91(4):771-786. doi: 10.1038/s41390-021-01497-4. Epub 2021 Apr 15. PMID 33859364
- [Background] Jazayeri Z, Sajadi M, Dalvand H, Zolfaghari M. Comparison of the effect of foot reflexology and body massage on physiological indicators and bilirubin levels in neonates under phototherapy. Complement Ther Med. 2021 Jun;59:102684. doi: 10.1016/j.ctim.2021.102684. Epub 2021 Feb 17. PMID 33609634
- [Background] Baniasadi H, Hosseini SS, Abdollahyar A, Sheikhbardsiri H. Effect of massage on behavioural responses of preterm infants in an educational hospital in Iran. J Reprod Infant Psychol. 2019 Jul;37(3):302-310. doi: 10.1080/02646838.2019.1578866. Epub 2019 Feb 21. PMID 30786750